CLINICAL TRIAL: NCT01158066
Title: Association Between NAFLD and Coronary Artery Calcification
Brief Title: Association Between Non-alcoholic Fatty Liver Disease (NAFLD) and Coronary Artery Calcification
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Liver Clinic, Ziv medical center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NAFLD and CAC
Record Dates: First submitted 2010-07-04; First posted 2010-07-08 (Estimated); Last update posted 2011-04-06 (Estimated); Status verified 2010-06

CONDITIONS: Coronary Artery Calcification
Keywords: NAFLD; Calcium score; Liver Fat; Visceral fat; excessive visceral fat; excessive liver fat accumulation; Biomarkers of insulin resistance (HOMA), inflammation (CRP) and (MDA-Paraoxonase)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CT cardiac (No Intervention): the patient will undergo cardiac CT
  Interventions: Procedure: CT Cardiac

INTERVENTIONS:
Procedure: CT Cardiac — the patient will undergo cardiac CT

SUMMARY:
Coronary artery disease are 8 times more prevalent in patients with NAFLD then the general population and are being considered the most common cause of death. Cardiac CT is a reliable non invasive method in demonstrating Coronary Plaques. However the association between coronary artery calcium score (CAC) and NAFLD remains controversial

DETAILED DESCRIPTION:
Coronary artery disease are 8 times more prevalent in patients with NAFLD that the general population and are being considered the most common cause of death. Cardiac CT is a reliable non invasive method in demonstrating Coronary Plaques. However the association between coronary artery calcium score (CAC) and NAFLD remains controversial. AIM: the aim is to evaluate the association between CAC score ( CT) and NAFLD (CT). the working hypothesis is that Beside the traditional risk factors including age, diabetes, NAFLD is also associated with moderate to high risk of CAD.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo cardiac CT for patients with low to intermediate risk for CAD

Exclusion Criteria:

* Patients with PCI or CABG will be excluded

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-01 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Total calcium score measurement | 1 month
  total calcium score will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- Ziv medical center liver unit, Safed, Israel, Israel